CLINICAL TRIAL: NCT05445050
Title: Development of Motion-Model Ultrasound Localization Microscopy to Support Breast Cancer Diagnosis and Therapy Monitoring in Patients
Brief Title: mULM to Support Breast Cancer Diagnosis and Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Elmar Stickeler, Univ.-Prof. Dr. med. Elmar Stickeler, RWTH Aachen University, RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 351-19; DRKS00023954 (Other: DRKS (German Clinical Trials Register))
Record Dates: First submitted 2022-05-27; First posted 2022-07-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Primary Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; ultrasound; microbubbles
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinical application of mULM to support breast cancer diagnosis and therapy (Other): The study arm includes three parts A, B and C. In part A, the scan protocol, including the injection of the clinically approved contrast agent SonoVue® and the data acquisition time range, is optimized based on the mULM measurements of participants with primary breast cancer.
  The following part B consists of 2D-mULM measurements applied to triple-negative breast cancer patients throughout their neoadjuvant chemotherapy cycles with the aim to evaluate to which degree 2D-mULM allows for an assessment of the tumor response during therapy.
  In the last part C, participants with neoplasms of uncertain dignity will be investigated by 2D- and 3D-mULM measurements and the accuracy of differentiation between the lesions assessed.
  Interventions: Diagnostic Test: Application and measurement of tumor vascularization using diagnostic contrast enhanced ultrasound (CEUS)

INTERVENTIONS:
Diagnostic Test: Application and measurement of tumor vascularization using diagnostic contrast enhanced ultrasound (CEUS) — Part A: performing CEUS with the contrast agent SonoVue® at two different doses and two different injection speeds in participants with primary breast cancer
  Part B: performing CEUS with the contrast agent SonoVue® using the established protocol from part A in participants undergoing neoadjuvant chemotherapy
  Part C: performing CEUS with the contrast agent SonoVue® using the established protocol from part A in participants with lesions of unknown dignity

SUMMARY:
The goal of this project is to adapt the super-resolution ultrasound imaging technology motion-model Ultrasound Localization Microscopy (mULM) to clinical application. In this exploratory patient study a scan protocol will be established to subsequently investigate whether mULM allows the assessment of the tumor response to neoadjuvant chemotherapy in participants with a primary breast cancer diagnosis as well as for the differentiation of benign and malignant breast tumors in participants with lesions of unknown dignity.

DETAILED DESCRIPTION:
This study on the clinical translation of the super-resolution ultrasound imaging technique motion-model ultrasound localization microscopy (mULM) is composed of three parts. First, an ultrasound scan protocol will be developed by providing patients with primary breast carcinoma with an ultrasound scan to assess the size, location, and structure of the tumor. Images in the form of B-mode ultrasound, elastography, and contrast ultrasound will be obtained, and mini-movies of the CEUS examinations will be evaluated in a post-processing step. There, individual microbubbles of the ultrasound contrast agent will be identified and tracked to reconstruct the microvasculature of the tumor lesions. Participants will each receive 2 different doses of the clinically approved ultrasound contrast agent SonoVue®. The morphological and functional parameters obtained through the post-processing with the mULM algorithm are then analyzed and subsequently validated with histological examinations. Finally, the ultrasound examination protocol will be optimized and the corresponding dosage of the ultrasound contrast agent determined.

The examination protocol established in the first section will subsequently be applied to patients with primary breast carcinoma receiving neoadjuvant chemotherapy. Contrast-enhanced ultrasonography will be performed at three time points during the chemotherapy cycles and will be performed to assess tumor perfusion through application of the mULM-algorithm. The dosage of contrast agent is based on the dosage found in the previous part of the study. The CEUS examination is followed by the infusion of the chemotherapeutic agent. After completion of neoadjuvant chemotherapy, surgical resection of the tumor and microscopic examination of the tissue are performed according to guidelines.

In the final part of the study, patients with suspected breast tumor lesions are examined. They will first receive non-contrast-enhanced diagnostic ultrasound (B-mode and elastography). A contrast-enhanced ultrasound examination is performed on the largest lesion. To further develop the mULM methodology, this is performed as both 2D and 3D acquisition. The dosage of the contrast agent examination is again based on the optimal dosage found in the first study part. This ultrasound procedure is followed by guideline-guided biopsy for histologic clarification of the tumors, assessing dignity, hormone receptor as well as and HER2/neu status, proliferation rate, and vessel density.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age ≥ 18 yrs
* histologically confirmed primary breast cancer including all intrinsic subtypes (study parts A and B)
* highly suspected primary breast cancer (study part C)
* treatment with neoadjuvant chemotherapy (study part B)
* persons who are legally competent and mentally able to follow the instructions of the study team

Exclusion Criteria:

* younger than 18 years
* hypersensitivity / allergy to sulfur hexafluoride, Macrogol 4000, distearoylphosphatidylcholine, dipalmitoylphosphatidylglycerol-sodium, palmitic acid
* right-left shunt,
* signs of cardiovascular instability
* acute endocarditis
* artificial heart valves
* acute systemic inflammation and/or sepsis
* overactive coagulation status and/or recent thromboembolic events
* end stage of liver and kidney diseases
* severe pulmonary hypertension (pulmonary arterial pressure > 90 mmHg)
* uncontrolled systemic hypertension
* acute respiratory distress syndrome
* pregnancy
* commitment of the patient to any resident institution by order of any court or authority
* expectation of missing compliance
* alcohol or drug abuse
* patients who are in a relationship of dependence or in a working relationship to the sponsor, the investigator or his representative

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Relative blood volume | Study Part A & C: approximately 1 day before surgical removal of tumor
  Relative blood volume in % - describes the degree of vascularization - measured with mULM
Blood flow | Study Part A & C: approximately 1 day before surgical removal of tumor
  Blood flow in mm/s - measured with mULM
Change of relative blood volume | Study Part B: at the beginning of (approximately 1 hour before) first, second and fourth cycle of neoadjuvant chemotherapeutic treatment (each cycle is 14 days)
  Change of relative blood volume in %
Change of blood flow | Study Part B: at the beginning of (approximately 1 hour before) first, second and fourth cycle of neoadjuvant chemotherapeutic treatment (each cycle is 14 days)
  Change of blood flow in mm/s

SECONDARY OUTCOMES:
Change of tumor size | Study Part B: at the beginning of (approximately 1 hour before) first, second and fourth cycle of neoadjuvant chemotherapeutic treatment (each cycle is 14 days)
  Change of tumor size determined based on ultrasound B-mode imaging

CONTACTS AND LOCATIONS:
Overall Officials: Elmar Stickeler, Prof Dr. med, Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- Department of Gynecology and Obstetrics Universitätsklinikum Aachen, AöR, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The study results will be published in at least one scientific article.